CLINICAL TRIAL: NCT02666924
Title: The Effects of Attending Language and Culturally Appropriate Cooking Classes on Glycemic Control, Diabetes Knowledge and Self-management in Chinese-Canadian Patients Living With Diabetes Mellitus Type Two: A Pilot Study
Brief Title: Cooking Classes for Chinese Canadian Patients Living With Diabetes
Acronym: CCDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, David E. Harris, MD, MD, FRCPC, Vancouver General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VCH RGH CCDS 1.1
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooking class (Experimental): The addition of diabetes cooking educational classes to standard diabetes education classes. Cooking classes are a series of four, four-hour sessions. These cooking classes will be led by a registered dietitian, a registered nurse and a chinese chef. Conducted in Mandarin or Cantonese. The cooking education focus is culturally specific teaching for Chinese-Canadian persons living with diabetes.
  Interventions: Dietary Supplement: Chinese-canadian specific cooking classes
- Control (Active Comparator): Type 2 diabetes educational classes, consisting of two sessions, one week apart, four-hour classes. These classes are taught by a registered dietitian and nurse, in Mandarin or Cantonese.
  Interventions: Other: Diabetes educational classes

INTERVENTIONS:
Dietary Supplement: Chinese-canadian specific cooking classes — Series of four, four-hour cooking classes, occurring monthly for four months. Each of the cooking classes in the series will have diabetes self-management learning objectives: food choices, meal planning and preparation, portion control, self-monitoring of blood glucose levels and physical activity.
  Arms: Cooking class
Other: Diabetes educational classes — Series of two, four-hour diabetes education classes, occurring weekly for two weeks. Each class is run by a registered dietitian and nurse, trained as clinical diabetes educators, as per standards of the canadian diabetes association. Classes include focused teaching of the background of diabetes, dietary recommendations for diabetes, lifestyle recommendations for diabetes, medications for diabetes, and general standard of living recommended for diabetes mellitus type 2.
  Arms: Control

SUMMARY:
This study aims to determine whether providing language and culturally appropriate cooking classes to Chinese Canadian individuals with diabetes will help to improve their diabetes control, knowledge and self care activities. The control group will receive current standard care of two diabetes education classes led by the dietitian and nurse. The intervention group will receive standard care and a series of four interactive cooking classes led by a dietitian, nurse and chef. We will compare the results of blood work, knowledge and self care questionnaires between the two groups to determine whether there are any benefits to attending these cooking classes.

DETAILED DESCRIPTION:
This is a study attempting to investigate whether a cooking class intervention will lead to improved glycemic control in Chinese-Canadian people in the community of Richmond, British Columbia. By providing culturally appropriate cooking classes, tailored to Chinese foods, culture and population, we will be able to address specific challenges that affect ethnic Chinese patients with diabetes living in Canada. This innovative program would serve to meet a need that is currently unmet in the community, by providing a hands-on opportunity for participants to try different foods, learn various culturally appropriate recipes, prepare meals together and learn how the foods being eaten affects blood glucose. These classes would also serve as an avenue to reinforce various diabetes self-management activities - including self-monitoring of blood glucose and the effects of physical activity. Also, participants may benefit from peer support and the sharing of experiences and advice with each other. Through this research study, we hope to demonstrate improved diabetes knowledge, self-care management and glycemic control for patients who attend the cooking classes.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in Type 2 Diabetes Education class in Mandarin or Cantonese at the Richmond Hospital Diabetes Education Centre.
2. Ability to understand and participate in all scheduled diabetes education classes and/or cooking classes;
3. Ability to complete the study questionnaires and standard of care glycemic bloodwork
4. Prior diagnosis of diabetes mellitus type 2
5. Persons who identify as chinese-canadian

Exclusion Criteria for this study includes:

1. Inability to provide informed consent;
2. Planned changes to diabetes medications during the study period, for example insulin titrations or oral medication adjustments;
3. Currently enrolled in another study involving interventions related to diabetes care and management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 6 months
  Change in Hemoglobin A1C

SECONDARY OUTCOMES:
Fasting lipid profile | 6 months
  Change in fasting lipid profile
Renal function | 6 months
  Change in Glomerular filtration rate
Albuminuria screen | 6 months
  Change in urinary Albumin to Creatinine ratio

OTHER OUTCOMES:
Diabetes self care activities | 3 months post intervention
  Summary of Diabetes Self-Care Activities Measure (SDSCA) model
Diabetes self knowledge assessment | 3 months post intervention
  Michigan Diabetes Knowledge Test

CONTACTS AND LOCATIONS:
Overall Officials: Graydon S Meneilly, MD, FRCPC, Study Director — UBC, Vancouver Coastal Health
Locations (1):
- Richmond Diabetes Education Center, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Mitchell S, Sahye-Pudaruth S, Blanco Mejia S, Chiavaroli L, Mirrahimi A, Ireland C, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Leiter LA, Josse RG. Effect of legumes as part of a low glycemic index diet on glycemic control and cardiovascular risk factors in type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1653-60. doi: 10.1001/2013.jamainternmed.70. PMID 23089999
- [Background] Chan YM, Molassiotis A. The relationship between diabetes knowledge and compliance among Chinese with non-insulin dependent diabetes mellitus in Hong Kong. J Adv Nurs. 1999 Aug;30(2):431-8. doi: 10.1046/j.1365-2648.1999.01098.x. PMID 10457246
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Yin Xu, Savage C, Toobert D, Wei Pan, Whitmer K. Adaptation and testing of instruments to measure diabetes self-management in people with type 2 diabetes in mainland China. J Transcult Nurs. 2008 Jul;19(3):234-42. doi: 10.1177/1043659608319239. PMID 18579863
- [Background] Fitzgerald JT, Funnell MM, Hess GE, Barr PA, Anderson RM, Hiss RG, Davis WK. The reliability and validity of a brief diabetes knowledge test. Diabetes Care. 1998 May;21(5):706-10. doi: 10.2337/diacare.21.5.706. PMID 9589228
- [Background] Fitzgerald JT, Funnell MM, Anderson RM, Nwankwo R, Stansfield RB, Piatt GA. Validation of the Revised Brief Diabetes Knowledge Test (DKT2). Diabetes Educ. 2016 Apr;42(2):178-87. doi: 10.1177/0145721715624968. Epub 2016 Jan 14. PMID 26769757